CLINICAL TRIAL: NCT07091045
Title: Effectiveness of Robot-Assisted Structured Foot-Ankle Sensorimotor Training in Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Esra TEKECİ, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-2627
Record Dates: First submitted 2025-07-09; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Robotic Rehabilitation; Virtual Reality Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-Assisted Foot-Ankle Training Protocol (REG): (Experimental): Stage 1: Vibration Training Applied for Proper Stepping on the Sole of the Foot and Proper Pressure Distribution: The first step of the training will be constant vibration, and the second step will be sensory localization training with vibration.
  Stage 2: Passive Joint Range of Motion Training with Virtual Reality: The platform will move the ankle passively (passive stretching).
  Stage 3: Joint Position Sense Training: The platform will bring the patient's ankle to a certain dorsiflexion position, the patient will be asked to feel and be aware of this angle, then the patient will be asked to return to the neutral position and perform ankle dorsiflexion at the angle that the platform initially brought.
  Stage 4: Active Joint Range of Motion Training with Virtual Reality: Along with active dorsiflexion, when necessary, assistance will be provided with the Assistance as Needed (AAN) control paradigm, a feature of the robotic device.
  Stage 5: It is the same as Stage 1
  Interventions: Other: Robot-Assisted Foot-Ankle Training
- Conventional Foot-Ankle Training Protocol (KEG): (Active Comparator): Stage 1: Sensory Training to the Sole of the Foot: In the first step of the training, the physiotherapist will manually apply constant pressure with a blunt object, and in the second step, sensory localization training with a blunt object will be performed.
  Stage 2: Passive Joint Range of Motion Training:
  The ankle will be manually moved passively (passive stretching) by the physiotherapist.
  Stage 3: Joint Position Sense Training: The physiotherapist will bring the patient's ankle to a certain dorsiflexion position, the patient will be asked to feel and be aware of this angle, then the patient will be asked to return to the neutral position and perform ankle dorsiflexion at the angle that the physiotherapist initially brought.
  Stage 4: Active Joint Range of Motion Training:
  This stage will be performed with manual assistance provided by the physiotherapist when necessary, along with active dorsiflexion.
  Stage 5: It is the same as Stage 1
  Interventions: Other: Conventional Foot-Ankle Training

INTERVENTIONS:
Other: Robot-Assisted Foot-Ankle Training — Stage 1: Vibration Training Applied for Proper Stepping on the Sole of the Foot and Proper Pressure Distribution: The first step of the training will be constant vibration, and the second step will be sensory localization training with vibration.
  Stage 2: Passive Joint Range of Motion Training with Virtual Reality: The platform will move the ankle passively (passive stretching).
  Stage 3: Joint Position Sense Training: The platform will bring the patient's ankle to a certain dorsiflexion position, the patient will be asked to feel and be aware of this angle, then the patient will be asked to return to the neutral position and perform ankle dorsiflexion at the angle that the platform initially brought.
  Stage 4: Active Joint Range of Motion Training with Virtual Reality: Along with active dorsiflexion, when necessary, assistance will be provided with the Assistance as Needed (AAN) control paradigm, a feature of the robotic device.
  Stage 5: It is the same as Stage 1
  Other Names: Robotic foot-ankle therapy in stroke
  Arms: Robot-Assisted Foot-Ankle Training Protocol (REG):
Other: Conventional Foot-Ankle Training — Stage 1: Sensory Training to the Sole of the Foot: In the first step of the training, the physiotherapist will manually apply constant pressure with a blunt object, and in the second step, sensory localization training with a blunt object will be performed. Stage 2: Passive Joint Range of Motion Training: The ankle will be manually moved passively (passive stretching) by the physiotherapist. Stage 3: Joint Position Sense Training: The physiotherapist will bring the patient's ankle to a certain dorsiflexion position, the patient will be asked to feel and be aware of this angle, then the patient will be asked to return to the neutral position and perform ankle dorsiflexion at the angle that the physiotherapist initially brought. Stage 4: Active Joint Range of Motion Training: This stage will be performed with manual assistance provided by the physiotherapist when necessary, along with active dorsiflexion. Stage 5: It is the same as Stage 1
  Arms: Conventional Foot-Ankle Training Protocol (KEG):

SUMMARY:
Stroke, one of the central nervous system (CNS) disorders, is a global public health problem due to its high mortality rate and level of physical and mental disability. It is the leading cause of death after heart disease and cancer and one of the most important causes of disability worldwide. After a stroke, motor and sensory disorders, activity and participation limitations and various complications related to these are observed in the lower extremities. As a result of these losses, balance, mobility and gait abnormalities lead to a decrease in quality of life and fall problems.

In recent years, the use of robot-assisted rehabilitation in physiotherapy has increased significantly with the support of engineering studies. Robotic and technology-supported trainings enable rehabilitation to be carried out at high intensity and repetition, treatment to be adapted according to the needs of the patient, patient exercise performance to be objectively monitored continuously, customized treatment protocols to be implemented and patients to be motivated with virtual reality technology.

Platform-based end effector robots used for ankle rehabilitation in the lower extremity after stroke allow active and passive joint range of motion training to be performed. In addition to such motor trainings, adding sensory (vibrotactile) localization and cognitive trainings to the treatment improves sensory-motor-cognitive integration.

In this context, with the proposed robot-assisted structured foot-ankle sensorimotor training protocol:

1. Vibration and sensory localization training applied for correct stepping on the sole of the foot (plantar) and correct pressure distribution,
2. Passive range of motion training supported by virtual reality,
3. Position sense training,
4. Active range of motion training supported by virtual reality and the "Assist-as-needed-AAN" control paradigm,
5. Vibration and sensory localization training applied for correct stepping on the sole of the foot (plantar) and correct pressure distribution, a holistic foot-ankle rehabilitation consisting of 5 stages of sensory-motor-cognitive training will be performed.

The aim of the project is to investigate the effectiveness of our structured training protocol, which includes sensory, motor and cognitive integration for foot-ankle rehabilitation, which we created with a robot-assisted foot-ankle system, in stroke patients. Our project aims to improve the tone, range of motion, joint position sense, walking performance, static and dynamic balance control, tactile perception levels and quality of life of the ankle movement and muscles (dorsiflexor and plantar flexor muscles) that are impaired after stroke. It is also aimed to bring a robot-assisted structured foot-ankle training protocol to the literature.

DETAILED DESCRIPTION:
Power analysis using G-Power version 3.1 yielded 90% power, a d=1.135 effect size, and a total sample size of n=30, with each group consisting of 15 observations. Participants will be randomly assigned to either the Robotic-Assisted Foot-Ankle Training Protocol (REG) or the Conventional Foot-Ankle Training Protocol (CEG). One group will receive training with the robotic foot-ankle platform, while the other group will receive conventional training (manual training with a physiotherapist). Exercise programs will last 6 weeks, 3 days a week, for 40-45 minutes. Progression will be provided using the AAN control paradigm on the robot, and by the physiotherapist in the conventional training.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 65 years,
* Ability to understand and follow study instructions,
* Ability to demonstrate coherent speech and spatial-temporal orientation skills, signed informed consent form,

  ≤ 2 ankle plantar flexor spasticity according to the Modified Ashworth Scale (MAS),
* Completion of all conventional physical therapy,
* Having had a stroke at least 6 months ago (individuals with chronic stroke),
* Ability to walk at least 10 m with or without any assistive device.

Exclusion Criteria:

* Cognitive impairment (Mini-Mental State Examination score ≤ 24),
* Having pathologies affecting walking or balance (orthopedic complications, lower extremity amputation, osteoporosis, etc.),
* Uncontrolled conditions (e.g. diabetes, hypertension, debilitating or immunosuppressive diseases),
* İmpairments affecting participants' ability to understand instructions,
* İnsufficient visual acuity to see a screen,
* Fixed or painful contractures of the paretic ankle.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (Tonus Assessment) | From enrollment to the end of treatment at 18 weeks
  The Modified Ashworth Scale (MAS) has six options: 0, 1, 1+, 2, 3, and 4. As the score increases, tone increases and the patient's condition worsens.
  Modified Ashworth Scale (MAS) Scores:
  0: No increase in muscle tone.
  1: Slight increase in muscle tone; felt as a sudden catch and release with minimal resistance at the end of the range of motion.
  1+: Slight increase in muscle tone; felt as a sudden catch followed by minimal resistance in less than half (<50%) of the remaining range of motion.
  2: More pronounced increase in muscle tone; felt throughout most of the range of motion, but the joint can be moved easily.
  3: Significant increase in muscle tone; passive movement is difficult. 4: Affected part(s) are rigid in flexion or extension.
Static balance assessment (Single Leg Stance Test) | From enrollment to the end of treatment at 18 weeks
  In the one-leg stance test, the patient is asked to stand on one leg without assistance, eyes open. The stopwatch is started the moment the patient's foot leaves contact with the ground. The stopwatch is stopped the moment the patient's foot touches the ground, and the time is recorded. The test will be repeated three times and the average calculated. Increasing single-leg standing time indicates progressive improvement.
Dynamic Balance Assessment (Timed up and Go Test) | From enrollment to the end of treatment at 18 weeks
  The TUG test, frequently used in stroke survivors, measures a participant's dynamic balance and walking ability by recording the time it takes to complete a series of tasks, including rising from a chair, walking 3 meters forward, turning 180°, and sitting back down. The test will be repeated three times and averaged.
  Individuals exceeding the upper age limit are at increased risk of falling. A walking speed greater than the upper limit of the range specified for their age group is associated with impaired performance.
Assessment of Joint Range of Motion (Electrogoniometer) | From enrollment to the end of treatment at 18 weeks
  Ankle ROM will be evaluated with an electrogoniometer. Ankle dorsi and plantar flexion ROM will be measured in the supine position. Eversion-inversion ROM will be measured in the prone position. An increase in ankle ROM will be considered positive in terms of progression.
Assessment of Joint Position Sense (electrogoniometer) | From enrollment to the end of treatment at 18 weeks
  Joint position sense is assessed using an electrogoniometer, first by passive positioning with eyes open, then by active repositioning with eyes open (passive and active repositioning, respectively). The physiotherapist will slowly and randomly move the ankle to three different dorsiflexion angles (e.g., 9°, 12°, 17°) determined based on the patient's ROM. The therapist will hold the ankle in each position for 5 seconds and ask the patient to memorize the ankle position. After the ankle is passively moved to the starting position, the patient will be asked to bring the ankle to the target point. Three different angles will be tested for each assessment, and the distance differences between the passively moved angles and the patient's moved points will be recorded. The test will be repeated three times and the average will be calculated. Increased ROM at these angles will be considered positive for progression.
Assessment of Walking Capacity (10 meter walking test) | From enrollment to the end of treatment at 18 weeks
  During the test, the patient walks at a normal walking speed between two markers 10 meters apart, and the total time elapsed is recorded in m/s. A decrease in walking time over the specified distance is considered positive for progression.
Assessment of Motor Performance (Fugl-Meyer Lower Extremity Assessment) | From enrollment to the end of treatment at 18 weeks
  It will be evaluated with the Fugl-Meyer Lower Extremity Assessment (FMA-LE). The FMA-LE examines hip, knee, and ankle movements, and hierarchical recovery is recorded from reflexive movements to synergistic and non-synergistic movements based on the Brunnstrom stage of recovery. The FMA-LE is a reliable parameter in patients with early, subacute, and chronic stroke.
  Classifications for severity of impairment have been proposed based on FMA Total Motor Scores (out of 100 points):
  < 50 = Severe 50-84 = Marked 85-94 = Moderate 95-99 = Mild
Assessment of Tactile Perception Levels (Semmes Weinstein Monofilament Test) | From enrollment to the end of treatment at 18 weeks
  The Semmes Weinstein Monofilament Test will be used. The test battery assesses sensory functions from light touch to pressure sensation by touching the subject with monofilaments ranging in thickness from 1.65 to 6.65.
  Classification for the SWM test:
  1.65-2.83 (green): normal sensation 3.22-3.61 (blue): diminished light touch sensation 3.84-4.31 (purple): diminished protective sensation 4.56-6.65 (red): loss of protective sensation 6.65 (no response): deep pressure perception.
Assessment of Quality of Life (Stroke Specific Quality of Life Scale-SSQOL) | From enrollment to the end of treatment at 18 weeks
  The Stroke-Specific Quality of Life (SS-QOL) scale is a patient-centered outcome measure intended to assess health-related quality of life (HRQOL) specific to stroke patients. Patients must answer each question on the SS-QOL with reference to the past week. It is a self-report measure containing 49 items across 12 domains: Mobility (6 items), Energy (3 items), Upper extremity function (5 items), Work/productivity (3 items), Mood (5 items), Self-care (5 items), Social roles (5 items), Family roles (3 items), Vision (3 items), Language (5 items), Thinking (3 items), and Personality (3 items).
  Completing the scale takes approximately 10-15 minutes. Items are rated on a 5-point Likert scale. There are three different response sets.
  Higher scores indicate better functioning. The SS-QOL provides both domain scores and an overall SS-QOL summary score. Domain scores are unweighted averages of the corresponding items, while the summary score is an unweighted average of all twelve domain score
Assessment of Satisfaction Level Related to the Robot (Quest Scale-Lıkert Scale-4's) | From enrollment to the end of treatment at 18 weeks
  Assessment of satisfaction with the robot: This will be assessed using a Quest-Likert scale. A 4-point Likert scale will be used for assessment. It is a survey methodology using four response options. Stroke patients express their level of satisfaction by selecting one of four options: 1 Strongly Disagree, 2 Disagree, 3 Agree, and 4 Strongly Agree. A higher score will be interpreted as increased satisfaction and positive patient progress.
Dynamic Balance Assessment (MiniBESTest) | From enrollment to the end of treatment at 18 weeks
  The Mini-BESTest, which has validity and reliability in assessing postural control and balance in individuals after stroke, consists of 14 items, each scored between 0 and 2, with a maximum score of 28. "0" indicates the lowest functional level and "2" indicates the highest functional level.
Assessment of Walking Capacity (2 minute walking test) | From enrollment to the end of treatment at 18 weeks
  The individual is encouraged to walk as fast as they can safely walk for 2 minutes without any assistance, and the test is administered between two cones set 15 meters apart. Data will be evaluated based on normative data for men and women, according to age groups. Increasing the distance walked over 2 minutes will be considered progressively more positive.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Medipol Üniversitesi, Istanbul, Istanbul
  - İstanbul Medipol Üniversitesi, Istanbul

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kwong PWH, Ng SSM, Chung RCK, Ng GYF. A structural equation model of the relationship between muscle strength, balance performance, walking endurance and community integration in stroke survivors. PLoS One. 2017 Oct 19;12(10):e0185807. doi: 10.1371/journal.pone.0185807. eCollection 2017. PMID 29049293
- [Background] Kim KH, Jang SH. Effects of Cognitive Sensory Motor Training on Lower Extremity Muscle Strength and Balance in Post Stroke Patients: A Randomized Controlled Study. Clin Pract. 2021 Sep 14;11(3):640-649. doi: 10.3390/clinpract11030079. PMID 34563008
- [Background] Kim H, Cho S, Lee H. Effects of passive Bi-axial ankle stretching while walking on uneven terrains in older adults with chronic stroke. J Biomech. 2019 May 24;89:57-64. doi: 10.1016/j.jbiomech.2019.04.014. Epub 2019 Apr 17. PMID 31060809
- [Background] Khalifeloo M, Naghdi S, Ansari NN, Akbari M, Jalaie S, Jannat D, Hasson S. A study on the immediate effects of plantar vibration on balance dysfunction in patients with stroke. J Exerc Rehabil. 2018 Apr 26;14(2):259-266. doi: 10.12965/jer.1836044.022. eCollection 2018 Apr. PMID 29740561
- [Background] Kavounoudias A, Roll R, Roll JP. The plantar sole is a 'dynamometric map' for human balance control. Neuroreport. 1998 Oct 5;9(14):3247-52. doi: 10.1097/00001756-199810050-00021. PMID 9831459
- [Background] de la Iglesia DH, Mendes AS, Gonzalez GV, Jimenez-Bravo DM, de Paz Santana JF. Connected Elbow Exoskeleton System for Rehabilitation Training Based on Virtual Reality and Context-Aware. Sensors (Basel). 2020 Feb 6;20(3):858. doi: 10.3390/s20030858. PMID 32041156
- [Background] Hussain I, Jany R. Interpreting Stroke-Impaired Electromyography Patterns through Explainable Artificial Intelligence. Sensors (Basel). 2024 Feb 21;24(5):1392. doi: 10.3390/s24051392. PMID 38474928
- [Background] Hoh JE, Semrau JA. The Role of Sensory Impairments on Recovery and Rehabilitation After Stroke. Curr Neurol Neurosci Rep. 2025 Mar 6;25(1):22. doi: 10.1007/s11910-025-01407-9. PMID 40047982
- [Background] Hesse S, Tomelleri C, Bardeleben A, Werner C, Waldner A. Robot-assisted practice of gait and stair climbing in nonambulatory stroke patients. J Rehabil Res Dev. 2012;49(4):613-22. doi: 10.1682/jrrd.2011.08.0142. PMID 22773263
- [Background] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721
- [Background] Forrester LW, Roy A, Krywonis A, Kehs G, Krebs HI, Macko RF. Modular ankle robotics training in early subacute stroke: a randomized controlled pilot study. Neurorehabil Neural Repair. 2014 Sep;28(7):678-87. doi: 10.1177/1545968314521004. Epub 2014 Feb 10. PMID 24515923
- [Background] Foley N, Murie-Fernandez M, Speechley M, Salter K, Sequeira K, Teasell R. Does the treatment of spastic equinovarus deformity following stroke with botulinum toxin increase gait velocity? A systematic review and meta-analysis. Eur J Neurol. 2010 Dec;17(12):1419-27. doi: 10.1111/j.1468-1331.2010.03084.x. PMID 20491885
- [Background] Ferry B, Compagnat M, Yonneau J, Bensoussan L, Moucheboeuf G, Muller F, Laborde B, Jossart A, David R, Magne J, Marais L, Daviet JC. Awakening the control of the ankle dorsiflexors in the post-stroke hemiplegic subject to improve walking activity and social participation: the WAKE (Walking Ankle isoKinetic Exercise) randomised, controlled trial. Trials. 2022 Aug 16;23(1):661. doi: 10.1186/s13063-022-06545-w. PMID 35974379
- [Background] Feigin VL, Brainin M, Norrving B, Martins S, Sacco RL, Hacke W, Fisher M, Pandian J, Lindsay P. World Stroke Organization (WSO): Global Stroke Fact Sheet 2022. Int J Stroke. 2022 Jan;17(1):18-29. doi: 10.1177/17474930211065917. PMID 34986727
- [Background] De Santis D, Zenzeri J, Casadio M, Masia L, Riva A, Morasso P, Squeri V. Robot-assisted training of the kinesthetic sense: enhancing proprioception after stroke. Front Hum Neurosci. 2015 Jan 5;8:1037. doi: 10.3389/fnhum.2014.01037. eCollection 2014. PMID 25601833
- [Background] Covaciu F, Pisla A, Iordan AE. Development of a Virtual Reality Simulator for an Intelligent Robotic System Used in Ankle Rehabilitation. Sensors (Basel). 2021 Feb 23;21(4):1537. doi: 10.3390/s21041537. PMID 33672161
- [Background] Cordo P, Lutsep H, Cordo L, Wright WG, Cacciatore T, Skoss R. Assisted movement with enhanced sensation (AMES): coupling motor and sensory to remediate motor deficits in chronic stroke patients. Neurorehabil Neural Repair. 2009 Jan;23(1):67-77. doi: 10.1177/1545968308317437. Epub 2008 Jul 21. PMID 18645190
- [Background] Cioni M, Esquenazi A, Hirai B. Effects of botulinum toxin-A on gait velocity, step length, and base of support of patients with dynamic equinovarus foot. Am J Phys Med Rehabil. 2006 Jul;85(7):600-6. doi: 10.1097/01.phm.0000223216.50068.bc. PMID 16788391
- [Background] Cho JE, Lee WH, Shin JH, Kim H. Effects of bi-axial ankle strengthening on muscle co-contraction during gait in chronic stroke patients: A randomized controlled pilot study. Gait Posture. 2021 Jun;87:177-183. doi: 10.1016/j.gaitpost.2021.04.011. Epub 2021 Apr 15. PMID 33945964
- [Background] Chen X, Liu F, Yan Z, Cheng S, Liu X, Li H, Li Z. Therapeutic effects of sensory input training on motor function rehabilitation after stroke. Medicine (Baltimore). 2018 Nov;97(48):e13387. doi: 10.1097/MD.0000000000013387. PMID 30508935
- [Background] Celletti C, Suppa A, Bianchini E, Lakin S, Toscano M, La Torre G, Di Piero V, Camerota F. Promoting post-stroke recovery through focal or whole body vibration: criticisms and prospects from a narrative review. Neurol Sci. 2020 Jan;41(1):11-24. doi: 10.1007/s10072-019-04047-3. Epub 2019 Aug 30. PMID 31468237
- [Background] Caldas R, Mundt M, Potthast W, Buarque de Lima Neto F, Markert B. A systematic review of gait analysis methods based on inertial sensors and adaptive algorithms. Gait Posture. 2017 Sep;57:204-210. doi: 10.1016/j.gaitpost.2017.06.019. Epub 2017 Jun 24. PMID 28666178
- [Background] Bouisset S, Do MC. Posture, dynamic stability, and voluntary movement. Neurophysiol Clin. 2008 Dec;38(6):345-62. doi: 10.1016/j.neucli.2008.10.001. Epub 2008 Oct 18. PMID 19026956
- [Background] Bonassi G, Biggio M, Bisio A, Ruggeri P, Bove M, Avanzino L. Provision of somatosensory inputs during motor imagery enhances learning-induced plasticity in human motor cortex. Sci Rep. 2017 Aug 24;7(1):9300. doi: 10.1038/s41598-017-09597-0. PMID 28839226
- [Background] Bensoussan L, Mesure S, Viton JM, Delarque A. Kinematic and kinetic asymmetries in hemiplegic patients' gait initiation patterns. J Rehabil Med. 2006 Sep;38(5):287-94. doi: 10.1080/16501970600694859. PMID 16931458
- [Background] Hakverdioglu Yont G, Khorshid L. Turkish version of the Stroke-Specific Quality of Life Scale. Int Nurs Rev. 2012 Jun;59(2):274-80. doi: 10.1111/j.1466-7657.2011.00962.x. Epub 2011 Nov 23. PMID 22591101
- [Background] Williams LS, Weinberger M, Harris LE, Clark DO, Biller J. Development of a stroke-specific quality of life scale. Stroke. 1999 Jul;30(7):1362-9. doi: 10.1161/01.str.30.7.1362. PMID 10390308
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Hosoi Y, Kamimoto T, Sakai K, Yamada M, Kawakami M. Estimation of minimal detectable change in the 10-meter walking test for patients with stroke: a study stratified by gait speed. Front Neurol. 2023 Jul 19;14:1219505. doi: 10.3389/fneur.2023.1219505. eCollection 2023. PMID 37538254
- [Background] Mahmoudzadeh A, Nakhostin Ansari N, Naghdi S, Sadeghi-Demneh E, Motamedzadeh O, Shaw BS, Shariat A, Shaw I. Effect of Ankle Plantar Flexor Spasticity Level on Balance in Patients With Stroke: Protocol for a Cross-Sectional Study. JMIR Res Protoc. 2020 Aug 21;9(8):e16045. doi: 10.2196/16045. PMID 32663137
- [Background] Bohannon, R. W. 2001. ''Measurement of joint range of motion in the rehabilitation of patients with stroke'', Stroke Rehabilitation, 22(4), 417-421.
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Perez-Cruzado D, Gonzalez-Sanchez M, Cuesta-Vargas AI. Parameterization and reliability of single-leg balance test assessed with inertial sensors in stroke survivors: a cross-sectional study. Biomed Eng Online. 2014 Aug 30;13:127. doi: 10.1186/1475-925X-13-127. PMID 25174611
- [Background] Harb A, Margetis K, Kishner S. Modified Ashworth Scale. 2025 Apr 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554572/ PMID 32119459
- [Background] Conforto AB, Ferreiro KN, Tomasi C, dos Santos RL, Moreira VL, Marie SK, Baltieri SC, Scaff M, Cohen LG. Effects of somatosensory stimulation on motor function after subacute stroke. Neurorehabil Neural Repair. 2010 Mar-Apr;24(3):263-72. doi: 10.1177/1545968309349946. Epub 2009 Nov 2. PMID 19884642
- [Background] Asin-Prieto G, Mercante S, Rojas R, Navas M, Gomez D, Toledo M, Martinez-Exposito A, Moreno JC. Post-stroke rehabilitation of the ankle joint with a low cost monoarticular ankle robotic exoskeleton: Preliminary results. Front Bioeng Biotechnol. 2022 Nov 25;10:1015201. doi: 10.3389/fbioe.2022.1015201. eCollection 2022. PMID 36507258
- [Background] Arene N, Hidler J. Understanding motor impairment in the paretic lower limb after a stroke: a review of the literature. Top Stroke Rehabil. 2009 Sep-Oct;16(5):346-56. doi: 10.1310/tsr1605-346. PMID 19903653
- [Background] An, S.H., Park, D-S., Limb, Ji-Y. 2017. ''Discriminative validity of the timed up and go test for community ambulation in persons with chronic stroke'', Phys Ther Rehabil Sci., 6 (4), 176-181
- [Background] Karimi-AhmadAbadi A, Naghdi S, Ansari NN, Fakhari Z, Khalifeloo M. A clinical single blind study to investigate the immediate effects of plantar vibration on balance in patients after stroke. J Bodyw Mov Ther. 2018 Apr;22(2):242-246. doi: 10.1016/j.jbmt.2017.04.013. Epub 2017 May 5. PMID 29861214
- [Background] http://dx.doi.org/10.1016/j.jbmt.2017.04.013